CLINICAL TRIAL: NCT05642689
Title: Evaluation of Iron Absorption From Ferric Ammonium Phosphate and Ferric Pyrophosphate From an Instant Milk Drink in Young Children
Brief Title: Evaluation of Fe Absorption From Iron Salt in Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: ETH Zurich (Switzerland) (Other); Food and Nutrition Research Institute, Philippines (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 09.07NRC
Record Dates: First submitted 2022-03-29; First posted 2022-12-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Double blind randomized crossover study with two parallel arms
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Other): Comparison of iron absorption from FAP to Ferrous sulfate in milk
  Interventions: Other: Iron fortified milk with iron salt labelled with 58Fe and 57Fe
- 2 (Other): Comparison of iron absorption from ferric pyrophosphate to Ferrous sulfate in milk
  Interventions: Other: Iron fortified milk with iron salt labelled with 58Fe and 57Fe

INTERVENTIONS:
Other: Iron fortified milk with iron salt labelled with 58Fe and 57Fe — Oral administration of a serving of iron labelled with stable isotope (2 mg Fe per serving) in 200ml of reconstituted milk once after a overnight fast. The alternate test drink was fed on the following day in the same fashion. The administration was repeated on day 3 and 4.
  Other Names: Iron fortified milk with ferrous ammonium posphate labelled with 57Fe; Iron fortified milk with ferrous sulfate labelled with 58Fe
  Arms: 1
Other: Iron fortified milk with iron salt labelled with 58Fe and 57Fe — Oral administration of a serving of iron labelled with stable isotope (2 mg Fe per serving) in 200ml of reconstituted milk once after a overnight fast. The alternate test drink was fed on the following day in the same fashion. The administration was repeated on day 3 and 4.
  Other Names: Iron fortified milk with ferrous sulfate labelled with 58Fe; Iron fortified milk with ferric pyrophosphate labelled with 57Fe
  Arms: 2

SUMMARY:
The primary objective was:

* to compare iron absorption in apparently healthy children aged 3-6y from an instant full cream milk drink fortified with ferric pyrophosphate or ferric ammonium phosphate relative to ferrous sulfate as the reference fortificant.
* To compare iron absorption from ferric pyrophosphate to ferric ammonium phosphate from the milk drink

ELIGIBILITY:
Inclusion Criteria:

* 3-6 years old (inclusive)
* Normal BMI for age (WHO standard)
* Apparently healthy, no metabolic or gastrointestinal disorder
* Non-anemic (WHO cut-off for respective age
* No medication or vitamin/mineral supplements will be consumed during the study
* Intake of Vitamin/mineral supplements will be discontinued 2 weeks before the start of the study
* Parents demonstrate an understanding of the given information and ability to comply with the study procedure
* Having obtained his/her parents or his/her legal representative's informed consent

Exclusion Criteria:

* With known gastrointestinal or metabolic disorder or experiencing significant blood losses over the past 6 months
* Possible to have medication during the study
* Currently participating or having participated another clinical trial during the past 3 months prior the beginning of this study
* Subject who cannot be expected to comply with treatment

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Determination of iron absorption from FAP and from ferric pyrophosphate relative to Ferrous sulfate | 14 days post isotope consumption
  It is based on calculated amount of 58Fe and 57Fe appearing in the blood. For that the shift of the iron isotope ratios in the blood samples collected 14 days after the last consumption of the last test drink are measured. The calculation of circulating iron is based on blood volume and hemoglobin concentration. For calculations of fractional absorption, 90% incorporation of the absorbed iron into red blood cells is assumed. The relative iron absorption from FAP and from ferric pyrophosphate relative to ferrous sulfate is then calculated as follows: Relative bioavailability of a salt (RBV %) = ( Fe absorption from an iron salt/ Fe absorption from ferrous sulfate)∗ 100. The comparison of the iron absorption from ferric pyrophosphate to that from ferric ammonium phosphate will be made by statistical analysis of data measured and calculated as described above.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walczyk T, Kastenmayer P, Storcksdieck Genannt Bonsmann S, Zeder C, Grathwohl D, Hurrell RF. Ferrous ammonium phosphate (FeNH(4)PO(4)) as a new food fortificant: iron bioavailability compared to ferrous sulfate and ferric pyrophosphate from an instant milk drink. Eur J Nutr. 2013 Jun;52(4):1361-8. doi: 10.1007/s00394-012-0445-y. Epub 2012 Sep 6. PMID 22956195